CLINICAL TRIAL: NCT01039415
Title: Attempts to Stop/Reduce Marijuana Among Dependent Users
Status: Completed | Type: Observational
Sponsor: University of Vermont (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, John Hughes, Professor of psychiatry, University of Vermont
Other Study IDs: CHRBS #09-005; R01DA024691 (NIH)
Record Dates: First submitted 2009-12-24; First posted 2009-12-25 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Marijuana Abuse; Marijuana Dependence
Keywords: marijuana; marijuana abuse; marijuana dependence; cannabis; substance-related disorder; abstinence
MeSH Terms: conditions — Marijuana Abuse; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to determine why and how marijuana users stop or reduce their marijuana use.

DETAILED DESCRIPTION:
The major aim of this study is to provide a better understanding of attempts to stop or reduce marijuana use that can be used to develop better behavioral treatments for marijuana dependence. The application will focus on adult daily marijuana users who try to stop or reduce their marijuana use in a real-world setting. Although prospective, natural history studies describing attempts to stop or reduce alcohol, heroin and tobacco use have proved useful, we know of no such study among adult marijuana users. Two pilot studies will develop measures and assess compliance with our procedures. The main study will recruit up to 400 adult marijuana smokers with the goal of a sample size of 200 participants with adequate compliance. Participants will call an Interactive Voice Recording (IVR) system daily for 3 months to report marijuana use, quit/reduction attempts, and events that might increase or decrease the probability of initiating a quit/reduction attempt or the success of an attempt. Follow-up at 6 months will track recent marijuana and other drug use. Knowing what motivates marijuana users to try to stop or reduce, and knowing which strategies for stopping marijuana use are successful, can help develop treatments for marijuana dependence. For example, if stopping tobacco when trying to stop marijuana decreases the chance of stopping marijuana, then smoking cessation should be done after stopping marijuana. Or if reducing marijuana often leads to cessation, then convincing those not interested in quitting marijuana to first try reducing may be helpful.

ELIGIBILITY:
Inclusion Criteria:

* daily marijuana smokers for at least 1 year

Exclusion Criteria:

* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adults 18 and older
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2010-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
initiation of a quit or reduction attempt | during 3 months of monitoring

SECONDARY OUTCOMES:
duration of a quit attempt | during the 3 months of monitoring

CONTACTS AND LOCATIONS:
Overall Officials: John Hughes, MD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States

REFERENCES:
- [Result] Hughes JR, Fingar JR, Budney AJ, Naud S, Helzer JE, Callas PW. Marijuana use and intoxication among daily users: an intensive longitudinal study. Addict Behav. 2014 Oct;39(10):1464-70. doi: 10.1016/j.addbeh.2014.05.024. Epub 2014 Jun 4. PMID 24935797
- [Result] Hughes JR, Naud S, Budney AJ, Fingar JR, Callas PW. Attempts to stop or reduce daily cannabis use: An intensive natural history study. Psychol Addict Behav. 2016 May;30(3):389-97. doi: 10.1037/adb0000155. Epub 2016 Feb 1. PMID 26828641
- [Result] Hughes JR, Naud S, Budney AJ, Fingar JR, Callas PW. Environmental cues and attempts to change in daily cannabis users: An intensive longitudinal study. Drug Alcohol Depend. 2016 Apr 1;161:15-20. doi: 10.1016/j.drugalcdep.2015.09.033. Epub 2016 Feb 6. PMID 26872879